CLINICAL TRIAL: NCT04413110
Title: PSG and Neuroendocrine Hormones in Subjective Cognitive Impaired Patients With Transformed Migraine
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University migraine
Record Dates: First submitted 2020-05-30; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Migraine
Keywords: MIGRAINE
MeSH Terms: conditions — Migraine Disorders | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-subjective cognitive impaired: Cases of migraine and non-subjective cognitive impaired
- Subjective cognitive impaired: Cases of migraine and subjective cognitive impaired
  Interventions: Device: Polysomnography
- Control group: Age and sex matched healthy controls
  Interventions: Device: Polysomnography

INTERVENTIONS:
Device: Polysomnography — PSG was carried out for 41 patients with subjective cognitive impairment and 41 age and sex-matched controls. PSG with standard EEG montage that includes bilateral EOG and four EEG leads were used. A single attended overnight PSG study was performed at the Clinical Neurophysiology Unit of Mansoura University Hospitals. Patients were studied in a quiet, darkened room with no medications were used to induce sleep. All participants underwent one night of laboratory-based PSG.
  Groups: Control group; Subjective cognitive impaired

SUMMARY:
Transformed migraine is the most common and challenging subtype of chronic daily headache disorders35. Patients with transformed migraine often report an evolutionary process that occurs over months or years in which headaches increase in frequency, change characteristics and ultimately result in patterns of daily or near-daily headaches resembling a mixture of tension-type headache and migraine.

DETAILED DESCRIPTION:
The present study aimed to investigate the presence and frequency of cognitive affection in patients with transformed migraines, as well as to analyze the association of cognitive affection with clinical features and headache impact, anxiety, depression, and quality of sleep.

ELIGIBILITY:
Inclusion Criteria:

-Patients included were adults with clinically confirmed of chronic migraine

Exclusion Criteria:

* Primary headache disorder other than migraine
* Secondary headache disorders other than medication-overuse headache or unclassified headache, or
* Aged under 18 years or older than 65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The diagnosis of headache disorders was based on the International Classification of Disease, Eleventh Revision (ICD-11). Patients included were adults with clinically confirmed of chronic migraine, completion of cognitive testing and questionnaires, and normal performance on cognitive tests based on normative data, stratified by gender, age, and education level.
Sampling Method: Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Polysomnography | 24-72 hours
  PSG was carried out for 41 patients with subjective cognitive impairment and 41 age and sex-matched controls. PSG with standard EEG montage that includes bilateral EOG and four EEG leads were used. A single attended overnight PSG study was performed at the Clinical Neurophysiology Unit of Mansoura University Hospitals. Patients were studied in a quiet, darkened room with no medications were used to induce sleep. All participants underwent one night of laboratory-based PSG.

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kavuk I, Yavuz A, Cetindere U, Agelink MW, Diener HC. Epidemiology of chronic daily headache. Eur J Med Res. 2003 Jun 30;8(6):236-40. PMID 12911872
- [Background] Bigal ME, Lipton RB, Tepper SJ, Rapoport AM, Sheftell FD. Primary chronic daily headache and its subtypes in adolescents and adults. Neurology. 2004 Sep 14;63(5):843-7. doi: 10.1212/01.wnl.0000137039.08724.18. PMID 15365134
- [Background] Silberstein SD. Chronic daily headache. J Am Osteopath Assoc. 2005 Apr;105(4 Suppl 2):23S-29S. PMID 15928350
- [Background] Bigal ME, Lipton RB. Modifiable risk factors for migraine progression. Headache. 2006 Oct;46(9):1334-43. doi: 10.1111/j.1526-4610.2006.00577.x. PMID 17040331
- [Background] Bigal ME, Lipton RB. Obesity is a risk factor for transformed migraine but not chronic tension-type headache. Neurology. 2006 Jul 25;67(2):252-7. doi: 10.1212/01.wnl.0000225052.35019.f9. PMID 16864817
- [Derived] Esmael A, Abdelsalam M, Shoukri A, Elsherif M. Subjective cognitive impairment in patients with transformed migraine and the associated psychological and sleep disturbances. Sleep Breath. 2021 Dec;25(4):2119-2126. doi: 10.1007/s11325-021-02308-0. Epub 2021 Feb 4. PMID 33543444